CLINICAL TRIAL: NCT02033824
Title: A Multicenter Prospective Randomized Clinical Trial Using Dehydrated Human Amnion/Chorion Membrane dHACM in Decompressive Craniectomy Patients to Reduce Postoperative Scarring
Brief Title: Amniotic Membrane in Decompressive Craniectomy to Reduce Scarring
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MiMedx Group, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AFCRAN001
Record Dates: First submitted 2013-11-21; First posted 2014-01-13 (Estimated); Last update posted 2018-08-23 (Actual); Status verified 2018-08

CONDITIONS: Scarring
MeSH Terms: conditions — Cicatrix | interventions — Craniotomy; Decompressive Craniectomy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 Control (Other): Will receive only traditional craniectomy
  Interventions: Procedure: Craniectomy
- Group 2 Treatment dHACM (Experimental): Will receive craniectomy, but with the addition of a piece of dHACM placed over any dural defect or dural closure.
  Interventions: Other: dHACM; Procedure: Craniectomy

INTERVENTIONS:
Other: dHACM — A piece of dHACM placed over any dural defect or dural closure during craniectomy.
  Other Names: AmnioFix®
  Arms: Group 2 Treatment dHACM
Procedure: Craniectomy — Removal of the skull flap followed by closure techniques per current SOC.
  Other Names: Decompressive Craniectomy

SUMMARY:
The purpose of this study is to evaluate the effectiveness of dHACM in reducing scar tissue formation in craniectomy patients as well as facilitating reoperation and repair. Specifically this study compares craniectomy without dHACM application to craniectomy with placement of dHACM between the galea and dura over dural suture line and/or exposed parenchyma.

ELIGIBILITY:
Inclusion Criteria:

* Adults ages 18 or older.
* Diagnosed with closed head trauma or cerebral infarction where decompressive craniectomy with durotomy is performed.
* Willingness to comply with study procedures.
* The patient's or legally authorized representative's (LAR's) ability to give full written consent.

Exclusion Criteria:

* Prior surgery at the site
* Participation in another ongoing trial
* Open cranial wounds
* Site exhibits clinical signs and symptoms of local infection.
* Current diagnosis of cancer at the site
* Prior radiation therapy treatment at the site.
* Patients on any investigational drug(s) or therapeutic device(s) within 30 days preceding screening.
* Known history of having Acquired Immunodeficiency Syndrome (AIDS) or HIV.
* Presence of any condition(s) which seriously compromises the subject's ability to complete this study, or has a known history of poor adherence with medical treatment.
* Currently taking medications which could affect graft incorporation (supervising physician's discretion).
* Allergy to gentamicin sulfate and/or streptomycin sulfate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2014-04; Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Degree of scarring between the galea and the dura, as assessed by the Ease of Dissection (EOD) Score and histological analysis upon reoperation in patients receiving craniectomy with durotomy. | 6 Months

SECONDARY OUTCOMES:
Intra- and post-operative complications at reoperation, as assessed by occurrence of violation of the dura and/or violation of the parenchyma. | 6 Months
Post-operative complications at original and re-operation | 6 Months
Peri-operative measures at original and re-operation | 6 Months
Survival | 6 Months

CONTACTS AND LOCATIONS:
Overall Officials: Chris Clare, MD, Principal Investigator — MiMedx Group, Inc.
Locations (2):
- United States (2):
  - Boulder Neurological Associates, Boulder, Colorado
  - Chattanooga Center for Neurological Research, Chattanooga, Tennessee